CLINICAL TRIAL: NCT06570850
Title: Efficacy of Colistin Monotherapy Versus Colistin Combined With Fosfomycin Against Carbapenem-Resistant Acinetobacter Baumannii Infections
Brief Title: Colistin Monotherapy vs Colsitin-fosfomycine in CRAB Infection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Parichat Salee, Assistant professor Parichat sales, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MED-2566-09378
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Infection Due to Carbapenem Resistant Acinetobacter
Keywords: carbapenem resistant Acinetobacter baumanni; CRAB; Colistin; Fosfomycin
MeSH Terms: interventions — colistinmethanesulfonic acid; Colistin; Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colistin group (Active Comparator): Participants receive intravenous colistin (colistinmethate soidum) 5 mg/kg/day (dosage will be adjusted according to creatinine clearance) and colistin nebulization at 80 mg every 8 hours in case of pneumonia.
  Interventions: Drug: Colistin Sodium Methanesulfonate
- Colistin plus fosfomycin group (Active Comparator): Participants receive intravenous colistin (colistinmethate soidum) (dosage regimen same as colistin group plus intravenous fosfomycin (dosage will be adjusted according to creatinine clearance and MIC).
  Interventions: Drug: Colistin Sodium Methanesulfonate plus Fosfomycin

INTERVENTIONS:
Drug: Colistin Sodium Methanesulfonate — Intravenous colistin (colistinmethate soidum) 5 mg/kg/day intravenous (dosage will be adjusted according to creatinine clearance). The duration of treatment ranges from 10 to 14 days, depending on the site of infection and clinical responsiveness.
  Other Names: Colistin
  Arms: Colistin group
Drug: Colistin Sodium Methanesulfonate plus Fosfomycin — Intravenous colistin(dosage is same as colistin group) plus intravenous fosfomycin(dosage will be adjusted according to MIC and creatinine clearance). The duration of treatment ranges from 10 to 14 days, depending on the site of infection and clinical responsiveness.
  Other Names: Colistin plus fosfomycin
  Arms: Colistin plus fosfomycin group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of colistin compared with colistin plus fosfomycin against carbapenem-resistant Acinetobacter baumanii infection in Thailand. The main questions it aims to answer the following main questions:

1. Which group has better clinical response at end of treatment
2. Which group has better clinical response at 72 hours and micrological cure at 72 hours and at end of treatment

DETAILED DESCRIPTION:
Participants will be randomized in a 1:1 ratio to receive a combination of intravenous colistin plus intravenous fosfomycin (combination group) or colistin alone (monotherapy group) to determine if monotherapy or combination therapy has a better outcome.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 20 years old patients who have CRAB infections (pneumonia, urinary tract infection, skin and soft tissue infection, bloodstream infection)
* Able to provide informed consent or having a legal proxy who can provide informed consent in case the subject is unable to provide consent on his own

Exclusion Criteria:

* Minimum inhibitory concentration (MIC) of colistin > 2 mg/L
* Complicated infection with inadequate source controlled
* Intracranial infection
* Infective endocarditis
* Intraabdominal infection
* Bone and joint infection
* Allergic to or have contraindication(s) to any treatment regimen in the study
* Polymicrobial infection with Carbapenem-resistant Psuedomonas aeruginosa, Carbapenem-resistant Enterobacterales (CRE), Vancomycin-resistant Enterococcus (VRE)
* Pregnancy
* Previous treatment with colistin or fosfomycin more than 96 hours
* Life expectancy of 24 hour or less
* Refusal to participate in the study
* Hospice treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with clinical response after completion of therapy | Baseline, day 10-14 (end of therapy)
  Clinical response are categorized as: clinical cure if participants recover all symptoms and signs of infection; partial response if they disappear only some of the initial symptoms and signs of infection, including the condition not fulfilling all the requirements for clinical cure; and clinical failure if participants have persistence or worsening of all symptoms and signs of infection despite antimicrobial treatment.

SECONDARY OUTCOMES:
Number of participants with clinical response at 72 hours of therapy | Baseline, day 3
  Clinical response are categorized as: clinical cure if participants recover all symptoms and signs of infection; partial response if they disappear only some of the initial symptoms and signs of infection, including the condition not fulfilling all the requirements for clinical cure; and clinical failure if participants have persistence or worsening of all symptoms and signs of infection despite antimicrobial treatment.
Number of participants with microbiological cure at 72 hours of therapy | Baseline, day 3
  Microbiological cure: no isolation of the causative agent in the infective site at 72 hours and end of treatment Microbiological failure: persistence of the causative agent in the infective site at 72 hours
Number of participants with microbiological cure after completion of therapy | Baseline, day 3
  Microbiological cure: no isolation of the causative agent in the infective site at 72 hours and end of treatment Microbiological failure: persistence of the causative agent in the infective site at 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Athitaya Luangnara, Principal Investigator — Chiang Mai University
Locations (1):
- Faculty of medicine, Chiang Mai university, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No